CLINICAL TRIAL: NCT01395992
Title: A Multicenter, Double-Blind, Fixed-Dose, Long-Term Extension Trial of the Safety of Asenapine in Subjects Diagnosed With Bipolar 1 Disorder Who Completed Protocol P05691 (Formerly 041044) (Phase3B, Protocol P05692 [Formerly 041045])
Brief Title: Long-Term Safety Extension Trial of Asenapine in Bipolar 1 Disorder Participants Who Completed Protocol P05691 (P05692)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05692; 2010-018410-78 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Bipolar I Disorder
MeSH Terms: interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine 5 mg (Experimental): Participants who were randomized to asenapine 5 mg twice per day (BID) during the P05691 study will be assigned to receive asenapine 5 mg BID on this extension study. Participant who were randomized to placebo during the P05691 study will be assigned to receive asenapine 5 mg BID on this extension trial.
  Interventions: Drug: asenapine
- Asenapine 10 mg (Experimental): Participants who were randomized to asenapine 10 mg BID during the P05691 study will be assigned to receive asenapine 10 mg BID on this extension study.
  Interventions: Drug: asenapine

INTERVENTIONS:
Drug: asenapine — asenapine 5 mg tablet, sublingually (SL) twice daily (BID) for 182 days
  Other Names: Saphris®, SCH 900274, Org 5222, Sycrest®
  Arms: Asenapine 5 mg
Drug: asenapine — asenapine 10 mg tablet, SL BID for 182 days
  Other Names: Saphris®, SCH 900274, Org 5222, Sycrest®
  Arms: Asenapine 10 mg

SUMMARY:
Participants who have completed the 3-week trial P05691 (NCT00764478) can be screened for eligibility for this 26-week extension study in which they will continue treatment. The primary purpose of this trial is to evaluate the long-term safety of asenapine.

ELIGIBILITY:
Inclusion criteria:

* Each participant must have completed the short-term trial P05691, and be judged by the investigator to likely benefit from continued treatment
* Each participant must have demonstrated an acceptable degree of compliance with trial medication, visits, and other requirements in the short-term trial P05691

Exclusion criteria:

* A participant must not have had any adverse event or other clinically significant finding(s) in the short-term trial P05691 that would prohibit the subject's continuation into this long-term extension trial
* A participant must not have any newly diagnosed or discovered psychiatric condition that would have excluded the subject from participation in the short-term trial P05691
* A participant must not be at imminent risk of self-harm or harm to others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing clinical and laboratory adverse events (AEs) | Baseline up to 212 days

CONTACTS AND LOCATIONS:
Locations (1):
- Forest Investigative Site 1000, Austin, Texas, United States